CLINICAL TRIAL: NCT05184114
Title: Clinical Significance of Subclinical Myocardial Involvement in Recovered COVID-19 Patients Using Cardiovascular Magnetic Resonance
Acronym: R-COVID-CMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ng Ming-Yen, Clinical Assistant Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UW 21-005
Record Dates: First submitted 2022-01-05; First posted 2022-01-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: COVID-19; Myocarditis
Keywords: COVID-19; Coronavirus; SARS-CoV-2; CMR; cardiac magnetic resonance imaging; Recovered COVID-19; Myocarditis
MeSH Terms: conditions — COVID-19; Myocarditis; Coronavirus Infections | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Recovered COVID-19 patients (Active Comparator): Recovered COVID-19 Patients will undergo three CMR examinations. The scans will take place at (i) within 2 weeks of confirmed recovery, (ii) 3 months after recovery and (iii) 1 year after recovery. At time of CMR examinations, patients will have blood tests.
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance, Blood Tests
- non-COVID-19 patients with viral respiratory infections (Experimental): non-COVID-19 Patients will undergo three CMR examinations. The scans will take place at (i) within 2 weeks of confirmed recovery, (ii) 3 months after recovery and (iii) 1 year after recovery. At time of CMR examinations, patients will have blood tests.
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance, Blood Tests
- Volunteers as age and gender matched controls. (Experimental): Volunteer controls will undergo one CMR examination. At time of CMR examinations, patients will have blood tests.
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance, Blood Tests
- Volunteers who planning to receive a 2-dose COVID-19 vaccine as vaccination controls (Experimental): Vaccination controls will undergo two CMR examinations. The scans will take place (i) within 2 weeks before received 1st dose of COVID-19 vaccine and (ii) within 2 weeks (preferably 5-7 days) after receiving the 2nd dose of COVID-19 vaccine. At time of CMR examinations, patients will have blood tests.
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance, Blood Tests

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance, Blood Tests — Imaging, blood investigations (white cell count, C-reactive protein, NT-proBNP, lactate dehydrogenase and high sensitivity troponin)

SUMMARY:
Introduction:

Coronavirus disease 2019 (COVID-19) remains a major health issue resulting in >800,000 deaths as of 30th August 2020. A concerning discovery of COVID-19 is the involvement of the myocardium. Several case studies including one from our group (recent study publication in JACC Cardiovascular Imaging led by the principal investigator of this grant application) have demonstrated subclinical myocardial inflammation in patients using cardiac magnetic resonance imaging (CMR) who have recovered from COVID-19. Furthermore at a cellular level, a recent autopsy study indicated that the severe acute respiratory syndrome coronavirus-2 is present in the myocardial tissue. The study further described invasion and viral progeny occurring in the myocardial interstitial cells and as such is a concerning development with the longer-term implications being unknown. These concerns have been noticed by the cardiology and non-cardiology medical community, with some expressing concerns of a new cause for cardiomyopathy and heart failure secondary to COVID-195. Therefore, it is critical that further studies are conducted to determine the longer-term outcome for patients.

DETAILED DESCRIPTION:
COVID-19 Cardiovascular Complications:

So far, COVID-19 has been linked to myocarditis, myocardial infarction, thrombosis/ hypercoaguable state and reduced cardiac function. At an early stage of the COVID-19 pandemic, it became apparent that cardiac complications were quite prevalent in COVID-19 patients, with a study from Wuhan showing 28% of patients having raised troponin levels and that raised troponin levels were correlated with poor outcome including death. In three case series using CMR to evaluate patients, the prevalence of myocardial infarcts ranged from 0% to 12%, myocardial inflammation was present in 56% to 60% of patients and reduced LV function was present in up to 7% of patients.

Role of CMR Imaging in COVID-19:

CMR is unique amongst the cardiac imaging modalities in providing a comprehensive evaluation of the heart structure, function and tissue characterisation. The European Society of Cardiology recognises CMR as the gold standard for assessing cardiac systolic function and volumes due to the high reproducibility between observers. Thus it allows for differences in cardiac systolic function and volumes to be detected earlier and with smaller sample sizes compared to echocardiography. CMR's tissue characterisation capabilities are unavailable to other modalities, and does not require ionising radiation or radioactive tracers (unlike computed tomography or nuclear imaging), which is ideal for follow-up testing. It has multiple techniques to identify myocardial inflammation / oedema (eg. T2/T1 mapping), focal fibrosis (eg. late gadolinium enhancement [LGE] quantification), and diffuse fibrosis (extracellular volume or ECV quantification). The newest pixel-wise quantitative T1/T2-mapping techniques are also named by the ESC as one of six most innovative technologies to evaluate patients with heart failure.

Thus, in the context of COVID-19, CMR is well positioned to assess for myocarditis and its long-term consequences, such as the development of myocardial fibrosis, cardiac remodeling and ultimately dysfunction and failure. This is attested to by the American College of Cardiology and European Society of Cardiology.

Knowledge Gap - Long-Term Impact of COVID-19 related Myocardial Inflammation:

Several studies have shown that for acute myocarditis, a majority of patients show a reduction in oedema and fibrosis, and improvement in left ventricular (LV) ejection fraction (LVEF). However, a proportion of patients show ongoing chronic myocarditis and deterioration on ventricular function, even progressing to dilated cardiomyopathy, clinical heart failure and death. The long-term impact of myocardial inflammation in COVID-19 patients is unknown. COVID-19 may follow a similar cardiac trajectory as other viral illnesses that affect the heart, and given the early reports of cardiac involvement post COVID-19, it is reasonable to expect that a proportion of COVID-19 survivors will develop adverse long-term consequences of cardiac morbidity and mortality. It is thus important to elucidate the determinants of clinical non-resolution of COVID-19 myocarditis, and to identify these signs early, before permanent damage occurs to cardiac structure and function. Furthermore, it is important to compare COVID-19 to patients with non-COVID-19 patients with viral respiratory infections to allow us to better understand the cardiovascular risks posed by COVID-19 compared to other viral respiratory illnesses.

Preliminary Data:

In addition to the aforementioned studies demonstrating myocardial involvement in COVID-19 survivors, our group has not only published similar findings in a CMR study, but concernedly, our patients had less severe (mild to moderate) initial COVID-19 and a majority were asymptomatic at follow-up, whilst the other studies were in patients with greater COVID-19 severity and had residual cardiac symptoms. Yet, the investigators still demonstrated that 56% of our cohort had imaging evidence of subclinical myocardial inflammation, a significant proportion of which also had serological markers (eg. troponin, c-reactive protein and white cell count) to support ongoing inflammation even at 2 months post hospital discharge. These findings are concerning in that many COVID-19 survivors have unrecognised myocardial inflammation that may be untreated, a proportion of which may resolve spontaneously, but some may go on to develop dilated cardiomyopathy and/or heart failure.

ELIGIBILITY:
Inclusion Criteria:

• Recovered COVID-19 patients

Definition of recovered COVID-19 patient:

* COVID-19 diagnosis = established by a positive reverse transcription polymerase chain reaction (RT-PCR) for severe acute respiratory syndrome coronavirus-2 [SARS-CoV2] and recovered from COVID-19.
* Recovery = based on two criteria: (1) two negative nasopharyngeal swab RT-PCR results >24 hours apart and (2) absence of fever and improvement in respiratory symptoms.

  * Recovered non-COVID-19 patients with viral respiratory infections confirmed with viral polymerase chain reaction testing AND with a confirmed negative COVID-19 RT-PCR test.
  * Age and gender matched controls with no cardiac risk factors, not on cardiac medications, no history of myocardial infarction, heart failure or myocarditis, negative COVID-19 RT-PCR test and negative COVID-19 antibodies test.
  * Vaccination controls who planning to receive a 2-dose COVID-19 vaccine, with no history of myocardial infarction, heart failure or myocarditis AND with a confirmed negative COVID-19 RT-PCR test.

Exclusion Criteria:

* Previous myocardial infarction or myocarditis unrelated to COVID-19 infection
* History of heart failure unrelated to COVID-19 infection
* Presence of pacemakers or implantable cardiac defibrillators
* Any contraindication for CMR testing
* Renal impairment with eGFR <45ml/min/1.73m2
* Limited life expectancy <1 year, for example due to pulmonary disease, cancer or significant hepatic failure
* Refusal or inability to sign an informed consent.
* Potential for non-compliance towards the requirements in the trial protocol (especially the medical treatment) or follow-up visits

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
The extent of myocardial involvement, as assessed by CMR tissue characterisation (T1/ T2/ ECV/ LGE), 2 weeks after patient recovery, at 3-months post discharge and at 1-year post discharge. | 1 year
The correlation of these myocardial characteristics to biventricular structure, function (CMR cine/strain), blood biomarkers of inflammation, clinical symptoms, and functional capacity (6 minute walk test) at all time-points | 2 years

SECONDARY OUTCOMES:
Number of Participants with followed-up beyond the end of this study to assess for hard outcomes such as death. | 2 years
Number of Participants with followed-up beyond the end of this study to assess for hard outcomes such as heart failure hospitalisation. | 2 years
Number of Participants with cardiac arrest. | 2 years
Number of Participants with ventricular tachycardia. | 2 years
Number of Participants with ventricular fibrillation. | 2 years
Rate of subclinical myocardial inflammation post COVID-19 vaccination. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng MY, Tam CH, Lee YP, Fong HTA, Wong CK, Ng WKC, Yeung MHY, Ling WI, Tsao S, Wan EYF, Ferreira V, Yan AT, Siu CW, Yiu KH, Hung IF. Post-COVID-19 vaccination myocarditis: a prospective cohort study pre and post vaccination using cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2023 Dec 7;25(1):74. doi: 10.1186/s12968-023-00985-2. PMID 38057820